CLINICAL TRIAL: NCT03612609
Title: Pilot Study to Detect DENGUE Virus in Sperm.
Acronym: DENGSPERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/18/0133; 2018-A01195-50 (Other: ID RCB)
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2019-08

CONDITIONS: Dengue
Keywords: Dengue virus; Semen
MeSH Terms: conditions — Dengue | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood, urine and semen sample (Other): 15 patients, with acute dengue virus infection and a positive RNA detection in blood or/and urines
  Interventions: Biological: blood, urine and semen sample

INTERVENTIONS:
Biological: blood, urine and semen sample — Men will give semen, urine and blood specimens 7 days after the beginning of clinical signs and 15, 30, 60 and 90 days after. Dengue virus RNA being diagnosed with blood and/or urine sample positive for dengue virus RNA. Dengue virus RNA will be detected in seminal plasma, native semen cells and processed spermatozoa.

SUMMARY:
The purpose of this study is to seek the presence of dengue virus in semen, to determine its localization and to assess the efficiency of spermatozoa processing methods to obtain virus free spermatozoa. This is a prospective study involving 15 patients, with acute dengue virus infection and a positive RNA detection in blood or/and urines. These results are important to understand the physiopathology of dengue virus infection and will help to counsel the infected patient in epidemic zona or returning from epidemic country. Moreover, they will help to define the management and viral safety procedures during Medically assisted Procreation in the context of dengue virus epidemic

DETAILED DESCRIPTION:
Dengue fever is a major cause of illness and death worldwide. The disease is caused by dengue virus (DENGV) which gets transmitted to humans by the bites of infected Aedes mosquitoes. The dengue virus is a flavivirus genus as for example the West Nile virus, yellow fever virus or Zika virus. In march 2018 a Dengue epidemic seems to start in La Reunion island.

dengue virus transmission occurs generally via the bite of the female mosquitoes while rare cases of non-vector transmission were reported. Only one case-report showed dengue virus in vaginal tract following dengue infection and any research was published about the links between male genital tract and dengue virus while a study revealed that 27 others viruses that can result in viremia have been found in human semen.

In this context, the purpose of this study is to seek the presence of dengue virus in semen, to determine its localization and to assess the efficiency of spermatozoa processing methods to obtain virus free spermatozoa.

This is a prospective study involving 15 patients, with acute dengue virus infection and a positive RNA detection in blood or/and urines. Men will give semen, urine and blood specimens 7 days after the beginning of clinical signs and 15, 30, 60 and 90 days after. Dengue virus RNA being diagnosed with blood and/or urine sample positive for dengue virus RNA. Dengue virus RNA will be detected in seminal plasma, native semen cells and processed spermatozoa. Semen sampling and processing will be performed within the ART laboratory of the University Hospital of La Reunion (St Pierre) and research of dengue virus RNA in the laboratory of Virology of Toulouse University Hospital. This study will identify the presence or absence of dengue virus seminal shedding, its dynamic, and in case of shedding, verify the efficiency of semen processing to obtain virus free spermatozoa.

These results are important to understand the physiopathology of dengue virus infection and will help to counsel the infected patient in epidemic zona or returning from epidemic country. Moreover, they will help to define the management and viral safety procedures during Medically assisted Procreation in the context of dengue virus epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Patient male aged 18 to 45 years
* Patient in acute phase of dengue virus infection and with clinical criteria (date of onset of known clinical signs) which if thet aren't specific can be highly evocative in an epidemic zone. For example: Fever, asthenia, rash, arthritis/arthralgia, myalgia, headache, conjunctivitis.
* Detection of the dengue virus genome by reverse transcriptase polymerase chain reaction in the blood or urine
* Patient who can move to the laboratory for samples
* Patient having given his free and informed consent and having signed the consent
* Patient affiliated with a social security scheme or equivalent

Exclusion Criteria:

* Patient with an ejaculation disorder or who cannot sperm collection or with a sperm volume abnormal (<1,5 ml).
* Patient under guardianship or under trusteeship
* Patient already included in a research protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
dengue virus genomic RNA in patient sperm | 6 month
  Search for presence of dengue virus genomic RNA in patients sperm when they are in the acute phase of the infection with reverse transcriptase polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bujan, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Saint-Pierre, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nedjadi T, El-Kafrawy S, Sohrab SS, Despres P, Damanhouri G, Azhar E. Tackling dengue fever: Current status and challenges. Virol J. 2015 Dec 9;12:212. doi: 10.1186/s12985-015-0444-8. PMID 26645066
- [Background] Horstick O, Martinez E, Guzman MG, Martin JL, Ranzinger SR. WHO dengue case classification 2009 and its usefulness in practice: an expert consensus in the Americas. Pathog Glob Health. 2015 Feb;109(1):19-25. doi: 10.1179/2047773215Y.0000000003. Epub 2015 Jan 28. PMID 25630344
- [Background] Horstick O, Tozan Y, Wilder-Smith A. Reviewing dengue: still a neglected tropical disease? PLoS Negl Trop Dis. 2015 Apr 30;9(4):e0003632. doi: 10.1371/journal.pntd.0003632. eCollection 2015 Apr. PMID 25928673
- [Background] Tomashek KM, Lorenzi OD, Andujar-Perez DA, Torres-Velasquez BC, Hunsperger EA, Munoz-Jordan JL, Perez-Padilla J, Rivera A, Gonzalez-Zeno GE, Sharp TM, Galloway RL, Glass Elrod M, Mathis DL, Oberste MS, Nix WA, Henderson E, McQuiston J, Singleton J, Kato C, Garcia Gubern C, Santiago-Rivera W, Cruz-Correa J, Muns-Sosa R, Ortiz-Rivera JD, Jimenez G, Galarza IE, Horiuchi K, Margolis HS, Alvarado LI. Clinical and epidemiologic characteristics of dengue and other etiologic agents among patients with acute febrile illness, Puerto Rico, 2012-2015. PLoS Negl Trop Dis. 2017 Sep 13;11(9):e0005859. doi: 10.1371/journal.pntd.0005859. eCollection 2017 Sep. PMID 28902845
- [Background] Chen R, Vasilakis N. Dengue--quo tu et quo vadis? Viruses. 2011 Sep;3(9):1562-608. doi: 10.3390/v3091562. Epub 2011 Sep 1. PMID 21994796
- [Result] Mons J, Mahe-Poiron D, Mansuy JM, Lheureux H, Nigon D, Moinard N, Hamdi S, Pasquier C, Dejucq-Rainsford N, Bujan L. Effects of Acute Dengue Infection on Sperm and Virus Clearance in Body Fluids of Men. Emerg Infect Dis. 2022 Jun;28(6):1146-1153. doi: 10.3201/eid2806.212317. PMID 35608553